CLINICAL TRIAL: NCT07129694
Title: A Randomized, Multicenter Study Comparing the Safety and Efficacy of CT-ACL001, a Regenerative Ligament, With Standard Treatment in Anterior Cruciate Ligament Reconstruction
Brief Title: Obtain Safety and Effectiveness of CT-ACL001, a Regenerative Ligament Using Biological Tissue, in ACLR
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: CoreTissue BioEngineering Inc. (Industry)
Collaborators: Japan Agency for Medical Research and Development (Other Government); Mediscience Planning, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CT-ACL001; jRCT2032240214 (Other: Japan Registry of Clinical Trials (jRCT))
Record Dates: First submitted 2025-05-12; First posted 2025-08-19 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Anterior Cruciate Ligament Rupture
Keywords: Anterior cruciate ligament reconstruction; Biological medical device; Regenerative ligament
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries | interventions — Anterior Cruciate Ligament Reconstruction

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Safety evaluation cohort; CT-ACL001 treatment group (Experimental): An acute safety evaluation group that will receive treatment with the test device without randomization: 7 cases
  Interventions: Device: Anterior cruciate ligament reconstruction
- Randomization cohort; CT-ACL001 treatment group (Experimental): Treatment with the test device (test device group): 38 cases
  Interventions: Device: Anterior cruciate ligament reconstruction
- Randomization cohort; autologous tendon treatment group (Active Comparator): Anterior cruciate ligament reconstruction with autologous tendon (knee flexor tendon) (control group): 19 cases
  Interventions: Procedure: Anterior cruciate ligament reconstruction

INTERVENTIONS:
Device: Anterior cruciate ligament reconstruction — Single-bundle anterior cruciate ligament reconstruction will be performed using the test device. In addition, single-bundle anterior cruciate ligament reconstruction will also be performed in the control group using autologous knee flexor tendons.
  Arms: Randomization cohort; CT-ACL001 treatment group; Safety evaluation cohort; CT-ACL001 treatment group
Procedure: Anterior cruciate ligament reconstruction — Single-bundle anterior cruciate ligament reconstruction will be performed using the test device. In addition, single-bundle anterior cruciate ligament reconstruction will also be performed in the control group using autologous knee flexor tendons.
  Arms: Randomization cohort; autologous tendon treatment group

SUMMARY:
A randomized, multicenter study comparing the safety and efficacy of CT-ACL001, a regenerative ligament, with standard treatment in anterior cruciate ligament reconstruction

DETAILED DESCRIPTION:
The study will target patients (18 years old or older and under 45 years old) who have suffered anterior cruciate ligament injuries that require reconstruction surgery, and will evaluate the safety and efficacy of the investigational device when used in reconstruction surgery, using patients who used autologous tendons (knee flexor tendons) as a comparison control.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18 years old or older and under 45 years old.
* Patients with anterior cruciate ligament injury who are candidates for reconstruction surgery.

Exclusion Criteria:

* Chronic anterior cruciate ligament injury (injury occurred more than 12 months ago).
* History of knee surgery, including anterior cruciate ligament surgery on the index side.
* Complication or history cruciate ligament injury on the opposite side, history of total knee arthroplasty, osteotomy around the knee, or osteosynthesis around the knee on the opposite side.
* Meniscus injury that requires extensive resection and is impossible to suture on the index side, collateral ligament injury or posterior cruciate ligament injury of 2° or more on the index side.
* Complication of osteoarthritis of the knee on the index side, KL classification 2° or higher.
* Complications of cartilage damage that cannot be treated by drilling or microfracture on the index side.
* Patients with infection in the index knee or inflammatory joint disease such as rheumatoid arthritis.
* Patients undergoing radiation therapy, chemotherapy, or both.
* Patients currently receiving treatment with systemic steroids, immunosuppressants, or both.
* Patients who are allergic to bovine products (e.g. meat).
* Patients who cannot discontinue returning to sports until 9 months after reconstruction surgery.
* Pregnant, breastfeeding and possibly pregnant patients.
* Female patients of childbearing potential and male patients who cannot agree to contraception for at least one year after reconstruction surgery.
* Patients who participated in other clinical trials within 4 weeks prior to reconstruction surgery.

Ages: 18 Years to 44 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 64 (Estimated)
Dates: Start 2024-11-25 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
Evaluation of IKDC Subjective Score using a dedicated evaluation form | 12 months after surgery
  The non-inferiority of the test device group to the control group will be evaluated 12 months after surgery using the IKDC Subjective Score.
  (maximum score: 100 and minimum score: 0, higher scores mean a better outcome)

SECONDARY OUTCOMES:
Measurement of Tibial Anterior Translation using a measuring device | 12 months after surgery
  Evaluate whether there is any significant difference in the amount of anterior tibial movement between the test device group and the comparison group 12 months after surgery.
Evaluation of Donor Site Morbidity using a dedicated evaluation form | 1 week, 1 month, 3 months and 6 months after surgery
  Donor site morbidity will be evaluated to determine whether the test device group is superior to the control group at 1 week, 1 month, 3 months, and 6 months after surgery.
  (maximum score: 96 and minimum score: 0, higher scores mean a better outcome)
Measurement of Knee Flexion Strength using a measuring device | 3 months, 6 months and 12 months after surgery
  In knee flexion strength evaluation (isometric knee flexion strength ratio of affected side: affected side/healthy side (%)), evaluate whether the affected side ratio is greater in the test device group than in the control group at 3 months, 6 months, and 12 months after surgery.
Evaluation of TEGNER-Activity-Score using a dedicated evaluation form | 6 months and 12 months after surgery
  Evaluate whether there are any significant differences in TEGNER-Activity-Scores between the test group and the comparison group at 6 and 12 months after surgery.
  (maximum score: 10 and minimum score: 0, higher scores mean a better outcome)
Incidence of additional surgery on the affected side | Through 12 months after surgery
  To evaluate whether there is a significant difference in the incidence (number) of additional surgeries on the affected side up to 12 months after surgery.
Graft rupture rate | Through 12 months after surgery
  Evaluate using MRI (T1, T2) to determine whether there is a significant difference in the graft rupture rate between the test device group and the comparison group up to 12 months after surgery.
Joint effusion | 1 month, 3 months and 6 months and 12 months after surgery
  Evaluate whether there is any significant difference between the test device group and the comparison group in the incidence of joint effusion requiring puncture (1 month after surgery, 3 months after surgery, 6 months after surgery, and 12 months after surgery).
Adverse events/malfunction rates | Through 12 months after surgery
  Evaluate all adverse events and malfunctions that occur after IC has been obtained and during the clinical trial period.

OTHER OUTCOMES:
Thigh Circumference | 1 week and 2weeks after surgery
  Regarding the thigh circumference on the affected side, the difference between pre-operative and post-operative measurements one week and two weeks after surgery will be evaluated to be smaller in the test device group compared to the control group.
Surgery time | At index procedure
  Evaluate whether the surgical time (test device group and comparison group) of the test device group was shorter than that of the comparison group when the same surgeon performed the surgery. The surgical time was defined as the time from the start of skin incision to the completion of all suturing.
Evaluation of IKDC Subjective Score using a dedicated evaluation form | 24 months after surgery
  Evaluate the non-inferiority of the test device group to the control group using the IKDC Subjective Score.
  (maximum score: 100 and minimum score: 0, higher scores mean a better outcome)
Incidence of additional surgery on the affected side | 24 months after surgery
  To assess whether there is a significant difference in the incidence (number) of additional surgeries on the affected side.
Graft rupture rate | 24 months after surgery
  MRI evaluation will reveal that there is no significant difference in graft rupture rate between the test device group and the comparison group.
Measurement of Tibial Anterior Translation using a measuring device | 24 months after surgery
  Evaluate whether there is any significant difference between the test device group and the comparison group in the amount of anterior tibial movement compared to the healthy side.
Measurement of Knee Flexion Strength using a measuring device | 24 months after surgery
  In knee flexion strength evaluation (isometric knee flexion strength ratio to affected side), it is evaluated that the test device group has a higher affected side ratio than the control group.
Evaluation of TEGNER-Activity-Score using a dedicated evaluation form | 24 months after surgery
  Evaluate whether there is no significant difference in the TEGNER-Activity-Scores between the test device group and the comparison group.
  (maximum score: 10 and minimum score: 0, higher scores mean a better outcome)

CONTACTS AND LOCATIONS:
Locations (6):
- Japan (6):
  - Hirosaki University Hospital, Hirosaki, Aomori
  - Hiroshima University Hospital, Hiroshima, Hiroshima
  - Hokkaido University Hospital, Sapporo, Hokkaido
  - Kobe University Hospital, Kobe, Hyōgo
  - Juntendo University Hospital, Bunkyo-ku, Tokyo
  - Tokyo Women's Medical University Hospital, Shinjuku-ku, Tokyo

IPD SHARING:
Plan to Share IPD: Undecided